CLINICAL TRIAL: NCT05734105
Title: An International, Phase 3, Randomized, Multicenter, Open-label Study of Ripretinib vs Sunitinib in Patients With Advanced GIST With KIT Exon 11 and Co-occurring KIT Exons 17 and/or 18 Mutations Who Were Previously Treated With Imatinib
Brief Title: A Study of Ripretinib vs Sunitinib in Patients With Advanced GIST With Specific KIT Exon Mutations Who Were Previously Treated With Imatinib
Acronym: INSIGHT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCC-2618-03-003; 2022-503058-37-00 (EU CTIS Number)
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: GIST
Keywords: advanced gastrointestinal tumors; gastrointestinal stromal tumors; imatinib; ripretinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ripretinib (Experimental): 150 mg QD of ripretinib (3×50 mg tablets) will be dosed continuously in repeated 42-day cycles.
  Interventions: Drug: Ripretinib
- Sunitinib (Active Comparator): 50 mg QD of sunitinib (4×12.5 mg capsules) will be dosed in 42-day cycles. Sunitinib will be given continuously for 4 weeks with a 2-week break.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Ripretinib — 50 mg tablets
  Other Names: QINLOCK, DCC-2618
  Arms: Ripretinib
Drug: Sunitinib — 12.5 mg tablets
  Other Names: Sutent
  Arms: Sunitinib

SUMMARY:
This is a Phase 3, 2-arm, randomized, open-label, global, multicenter study comparing the efficacy of ripretinib to sunitinib in participants with GIST who progressed on first-line treatment with imatinib, harbor co-occurring KIT exons 11+17/18 mutations, and are without KIT exon 9, 13, or 14 mutations. Upon disease progression as determined by an independent radiologic review, participants randomized to sunitinib will be given the option to either crossover to receive ripretinib 150 mg QD or discontinue sunitinib.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Histologic diagnosis of GIST with co-occurring KIT exons 11+17/18 mutations confirmed by ctDNA sample.
3. Participants must have advanced GIST and radiologic progression on imatinib treatment.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤2 at screening.
5. Female participants of childbearing potential must have a negative pregnancy test at screening and prior to the first dose of study drug.
6. Participants of reproductive potential must agree to follow contraception requirements.
7. Participants must have at least 1 measurable lesion according to mRECIST v1.1 within 21 days prior to the first dose of study drug.
8. Adequate organ function and bone marrow reserve based on laboratory assessments performed at screening.

Exclusion Criteria:

1. History of KIT exon 9 mutation or detection of KIT exon 9, 13, or 14 mutations in a ctDNA sample.
2. Has known active central nervous system metastases.
3. New York Heart Association Class II-IV heart disease, myocardial infarction within 6 months of Cycle 1 Day 1, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension, or congestive heart failure.
4. Use of strong or moderate inhibitors or inducers of cytochrome P450 (CYP) 3A prior to the first dose of study drug, and consumption of grapefruit or grapefruit juice within 14 days prior to the first dose of study drug.
5. Major surgeries (eg, abdominal laparotomy) within 4 weeks of the first dose of study drug.
6. Known human immunodeficiency virus or hepatitis C infection only if the participant is taking medications that are excluded per protocol, acute or chronic hepatitis B, or acute or chronic hepatitis C infection.
7. Gastrointestinal abnormalities including, but not limited to:

   1. inability to take oral medication
   2. malabsorption syndromes
   3. requirement for intravenous alimentation
8. Any active bleeding excluding hemorrhoidal or gum bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to end of treatment; up to approximately 48 months
  The time from randomization until documented progressive disease (PD) based on IRR per mRECIST or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to end of treatment; up to approximately 48 months
  Compare ORR by IRR of ripretinib vs sunitinib using mRECIST
Overall Survival (OS) | Up to approximately 48 months
  Compare OS of ripretinib vs sunitinib

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team, Study Director — Deciphera Pharmaceuticals, LLC
Locations (70):
- United States (20):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Northwell Health Cancer Institute/ R.J. Zuckerberg Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (2):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Alfred Health, Melbourne, Victoria
- Brazil (6):
  - INCA - Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro
  - CEPEN - Centro de Pesquisa e Ensino em Saude de Santa Catarina, Florianópolis, Santa Catarina
  - Hospital de Cancer de Barretos - Fundacao Pio XII, Barretos, São Paulo
  - Hospital Sirio-Libanes, São Paulo, São Paulo
  - Hospital 9 de Julho, São Paulo, São Paulo
  - AC Camargo Câncer Center, São Paulo, São Paulo
- Canada (4):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Chile (2):
  - Clínica San Carlos De Apoquindo Red Salud UC Christus, Las Condes, RM
  - Centro de Oncología de Precisión, Santiago, RM
- France (5):
  - CHU Dijon, Dijon, Bourgogone
  - Centre Eugène Marquis, Rennes, Ille et Vilaine
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Helios Klinikum Berlin-Buch, Berlin
  - University Hospital Essen (Universitätsklinikum Essen), Essen
  - Heidelberg University Hospital, Heidelberg
  - Universitares Krebszentrum Leipzig, Leipzig
- Italy (7):
  - Istituto Nazionale Tumori IRCCS Fondazione "G Pascale", Naples, Napoli
  - U.O.C. Oncologia Medica, Palermo, Palermo
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Oncologico Veneto-IOV IRCCS, Padua
  - Università Campus Bio-Medico di Roma, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano
- Netherlands (2):
  - UMC Groningen, Groningen
  - LUMC, Leiden
- Oslo University Hospital, Oslo, Norway, Norway
- Narodowy Instytut Onkologii Im . Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw, Warszawa, Poland
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital Universitario Vall d'Hebron, Barcelona, Barcelona
  - Complejo Hospitalario Universitario de Vigo - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Instituto Valenciano de Oncologia - IVO, Valencia, Valencia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Centra de Asturias, Oviedo
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (2):
  - The Royal Marsden Hospital NHS Foundation Trust, London, Greater London
  - St. James University Hospital, Leeds, West Yorkshire

REFERENCES:
- [Derived] George S, Blay JY, Chi P, Jones RL, Serrano C, Somaiah N, Gelderblom H, Zalcberg JR, Reichmann W, Sprott K, Cox P, Sherman ML, Ruiz-Soto R, Heinrich MC, Bauer S. The INSIGHT study: a randomized, Phase III study of ripretinib versus sunitinib for advanced gastrointestinal stromal tumor with KIT exon 11 + 17/18 mutations. Future Oncol. 2024;20(27):1973-1982. doi: 10.1080/14796694.2024.2376521. Epub 2024 Sep 4. PMID 39229786
- See also: INSIGHT Patient Website — https://www.exploreinsightgist.com/
- See also: INSIGHT Physician Website — https://www.theinsightgiststudy.com/en-US